CLINICAL TRIAL: NCT01486745
Title: Is There a Role for Using NMR Urine Metabolomics as a New Method of Screening for Colorectal Cancer?
Brief Title: Urine Metabolomics and Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: MTI-2008; 514 (Other: U of A HREB)
Record Dates: First submitted 2011-12-03; First posted 2011-12-06 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Colorectal Polyps
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal colonoscopy
- Colonic polyps
- Colorectal cancer patients
- Breast & Prostate Cancer patients

SUMMARY:
This is a prospective, multi-centered study to assess whether urine metabolomics can play a role in the screening of colorectal cancer (CRC). Urine samples will be collected from 1000 patients going through an established CRC screening program, and from a further 500 patients who already have a diagnosis of CRC. Using nuclear magnetic resonance (NMR) spectroscopy, the 1H NMR spectrum of urine samples will be analyzed for specific metabolites, and establish the metabolomic signature of colorectal cancer. The results from metabolomic urinalysis of this screening cohort will be compared with results from colonoscopy, histological descriptions, fecal occult blood testing (FOBT), and fecal immune testing (FIT) to assess the accuracy of urine metabolomics in identifying patients with polyps and malignancies. The urine metabolomic results from the colorectal cancer group will be correlated with operative, histological and clinical staging to define the role of urine metabolomics in assessing colorectal cancer type, location and stage. Additionally approximately 300 urine samples from breast cancer patients and 300 from prostate cancer patients will be collected to validate that the colorectal cancer signature is unique.

ELIGIBILITY:
Inclusion Criteria:

For Screening group (normal colonoscopy & colonic polyps):

* asymptomatic, 50-75 year old, without personal or family history of CRC/polyps
* asymptomatic, 40-75 year old, known personal or first-degree family history of either CRC or polyps

For Cancer group:

* any patient with diagnosis of colorectal cancer
* any patient with diagnosis of prostate cancer
* any patient with diagnosis of breast cancer

Exclusion Criteria:

For screening group:

* hematochezia
* inflammatory bowel disease
* on anticoagulation for reasons other than atrial fibrillation
* significant co-morbidities

For Cancer group:

* already had neoadjuvant treatment at time of urine collection
* no invasive cancer at time of urine collection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing colorectal cancer screening Patients with diagnosis of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 2175 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haili Wang, MD FRCS(C), Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Eisner R, Greiner R, Tso V, Wang H, Fedorak RN. A machine-learned predictor of colonic polyps based on urinary metabolomics. Biomed Res Int. 2013;2013:303982. doi: 10.1155/2013/303982. Epub 2013 Nov 7. PMID 24307992